CLINICAL TRIAL: NCT06800443
Title: A Cosmetic Study to Measure the Change in Tooth Colour After Using Instant Whitening Prototypes Compared to a Negative Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ORL-WHI-3378
Record Dates: First submitted 2025-01-13; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Tooth Color
MeSH Terms: interventions — Charcoal; blue covarine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Test toothpaste 1 (Experimental): Silica-based toothpaste containing charcoal, clay, blue covarine, green covarine and fluoride as sodium fluoride
  Interventions: Other: Silica-based fluoride toothpaste containing clay, charcoal, blue covarine and green covarine
- Test toothpaste 2 (Experimental): Silica-based toothpaste containing blue covarine and fluoride as sodium monofluorophosphate
  Interventions: Other: Silica-based fluoride toothpaste with blue covarine
- Test toothpaste 3 (Experimental): Silica-based toothpaste containing blue covarine and fluoride as sodium monofluorophosphate
  Interventions: Other: Silica-based fluoride toothpaste with blue covarine
- Control toothpaste (Other): Control silica-based toothpaste containing fluoride as sodium fluoride
  Interventions: Other: Control silica-based fluoride toothpaste

INTERVENTIONS:
Other: Silica-based fluoride toothpaste containing clay, charcoal, blue covarine and green covarine — Silica-based toothpaste containing charcoal, clay, blue covarine, green covarine and fluoride as sodium fluoride
  Arms: Test toothpaste 1
Other: Silica-based fluoride toothpaste with blue covarine — Silica-based toothpaste containing lower level of blue covarine and fluoride as sodium monofluorophosphate
  Arms: Test toothpaste 2
Other: Silica-based fluoride toothpaste with blue covarine — Silica-based toothpaste containing higher level blue covarine and fluoride as sodium monofluorophosphate
  Arms: Test toothpaste 3
Other: Control silica-based fluoride toothpaste — Control silica-based toothpaste containing fluoride as sodium fluoride
  Arms: Control toothpaste

SUMMARY:
This will be a double blind, randomised, four-group crossover study. This study will involve 5 visits to the study site, with a wash-out period of 1 week between visits. Visit 1 will be for screening, participants who meet inclusion and exclusion criteria (including having Vita shade score of 2M2, 3R1.5, 2R2.5, 3L1.5, 2L2.5, 4M1, 2M3, 3M2, 4R1.5, 4L1.5, 3L2.5, 3R2.5, 5M1, 4M2, 3M3 from VITA 3D-MASTER Shade Guide) will be accepted onto the study. At each test visit (visit 2 - 5), participants will have images taken of their front upper incisors using a a Video-based Digital Imaging System (VDIS) pre- and post-brushing with randomly allocated test or control toothpaste [1.5g for 90 seconds, followed by water rinse]. The digital images will be analysed using the VDIS image analysis software and the mean CIELAB and WIO of the upper central incisors will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Two upper central incisors must be natural.
* The two upper central incisors must be within the colours of 2M2, 3R1.5, 2R2.5, 3L1.5, 2L2.5, 4M1, 2M3, 3M2, 4R1.5, 4L1.5, 3L2.5, 3R2.5, 5M1, 4M2, 3M3 from VITA 3D-MASTER Shade Guide.
* The two upper central incisors must be free of intrinsic stain e.g. caused by tetracycline, fluorosis etc.
* The two upper central incisors must be extrinsic stain free.
* Willing to sign an informed consent form and complete a medical history questionnaire.

Exclusion Criteria:

* Two upper central incisors have any caps, crowns, veneers or cracks in the teeth, have excessive gum recession, or have restorations on the distal, mesial, buccal, incisor edge in the opinion of the dentist and technician.
* Smoker (including e-cigarettes) or chews tobacco.
* Are diabetic
* Currently pregnant or breast feeding.
* Currently having orthodontics bands, partial removable dentures.
* Currently experiencing severe oral problems such as untreated caries, gingivitis or periodontal disease.
* Regular use of medication, which in the opinion of the study dentist, could interfere with study objectives.
* Known allergies to the toothpaste ingredients or to any dental materials.
* Use of tooth bleaching products in the past 6 months.
* Have been using whitening oral care products in the last 12 weeks or had a scale and polish in the last 3 months.
* Have or have had a medical condition that in the opinion of the study dentist would make them unsuitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2019-01-04 (Actual); Study Completion 2019-01-04 (Actual)

PRIMARY OUTCOMES:
Tooth whiteness index (WIO) (average value from two upper central incisors | Immediately after brushing
  Digital images of the upper central incisors will be taken before and immediately after brushing with toothpaste using a Video-based Digital Imaging System (VDIS). WIO will be obtained from VDIS images[1]. The outcome measure per participant will be the average values from two upper central incisor teeth. Increase in WIO means whiter.
  [1] Luo, Wen et al. J Dent. 2017;67S:S15-S19.

SECONDARY OUTCOMES:
Tooth Color Lightness L* (average value from two upper central incisors) | Immediately after brushing
  Digital images of the upper central incisors will be taken before and immediately after brushing with toothpaste using a Video-based Digital Imaging System (VDIS). L* will be obtained from VDIS images[1]. L* (Lightness) is one of the axes in CIELAB 3D color space. L* axis runs vertically and represents the lightness of the color. It ranges from 0 (black) to 100 (white). An increase in L* indicates tooth is lighter in color.
  [1] Luo, Wen et al. J Dent. 2017;67S:S15-S19.
Tooth Color a* (red/green) (average value of two upper central incisors) | Immediately after brushing
  Digital images of the upper central incisors will be taken before and immediately after brushing with toothpaste using a Video-based Digital Imaging System (VDIS). a* will be obtained from VDIS images[1]. a* (red-green) is one of the axes in CIELAB 3D color space. a* axis runs horizontally and represents the color's position between red and green. Positive values indicate a shift towards red, while negative values indicate a shift towards green.
  [1] Luo, Wen et al. J Dent. 2017;67S:S15-S19.
Tooth Color b* (blue/yellow) (average of two upper central incisors) | Immediately after brushing
  Digital images of the upper central incisors will be taken before and immediately after brushing with toothpaste using a Video-based Digital Imaging System (VDIS). b* will be obtained from VDIS images[1]. b* (blue-yellow) is one of the axes in CIELAB 3D color space. The b* axis runs horizontally and represents the color's position between blue and yellow. Positive values indicate a shift towards yellow, while negative values indicate a shift towards blue.
  [1] Luo, Wen et al. J Dent. 2017;67S:S15-S19.

CONTACTS AND LOCATIONS:
Locations (1):
- SPRIM China, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
Participant consent not available for this type of sharing.

REFERENCES:
- [Derived] Zhang L, Joiner A, Gupta AK, Barili M, Platten S, McDonald MD, Luo W, Matheson JR. Effect of Blue Covarine Toothpastes on Tooth Colour: A Randomised Crossover Study. Int Dent J. 2025 Oct;75(5):100938. doi: 10.1016/j.identj.2025.100938. Epub 2025 Aug 19. PMID 40834827